CLINICAL TRIAL: NCT02231151
Title: Providing Visual Feedback of Quality of CPR During Pediatric Cardiac Arrest: Does Point of View Matter?
Brief Title: Visual Feedback of CPR: Does Point of View Matter?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KidSIM Simulation Program (Network)
Responsible Party: Principal Investigator, Nicola Robertson, KidSim Aspire Coordinator, KidSIM Simulation Program
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: CPR Point of View
Record Dates: First submitted 2014-08-22; First posted 2014-09-04 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: CPR Quality Assessment
Keywords: CPR quality assessment; Visual CPR assessment; Position relative to patient

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pediatric Acute Care Professionals (Experimental): Individuals must work in ER or ICU setting regularly or rotate through this setting with up to date BLS/PALS/ACLS certification. The participants will be required to rate the CPR based on accuracy for each video shown. The type of CPR error(s) shown to the individuals will be randomized.
  Interventions: Behavioral: The type of CPR error(s) shown to the individual

INTERVENTIONS:
Behavioral: The type of CPR error(s) shown to the individual — Participants will be randomly assigned 12 videos to watch and rate the CPR quality of each. Investigators will be blind to the identity of the participants.

SUMMARY:
The investigators will look at how accurate pediatric healthcare workers are at judging quality of Cardiopulmonary Resuscitation, by observation of the chest compressions, and if they are more accurate at a certain position near the patient. The investigators will do this by having participants fill out a survey about the quality of the Cardiopulmonary Resuscitation in several recorded resuscitation scenarios.

DETAILED DESCRIPTION:
Pediatric cardiac arrest leads to significant productive years lost, and has a huge emotional impact on families and caregivers. High quality CPR is the most important predictor for outcome in cardiac arrest. Human visual observation is commonly used and important to evaluate CPR quality. Interestingly, the accuracy of healthcare providers' visual assessment of CPR quality is unknown.

Primary Objective: To determine the accuracy of visual CPR assessment. Secondary Objective: 1) To identify the optimal position relative to the patient for accurate CPR assessment. 2) To determine health care practitioners' accuracy in identifying CPR errors.

Methods: We will videotape both good quality CPR and poor quality CPR in a simulated resuscitation. We will record 4 videos, one depicting high quality CPR, and 3 depicting the most common mistakes made when performing chest compressions, and these will be videotaped from the foot, head and side of the patient. Pediatric acute care professionals will be recruited to watch a randomized set of all 12 video clips, and fill out a brief and simple questionnaire on their assessment of the quality of the CPR being performed.

To assess the accuracy of the CPR quality, quantitative data on the quality of the CPR being performed during each of the 4 videotaped events will be captured and confirmed using a Laerdal CPRcard© (depth and rate) and the paediatric simulator SimJr© (recoil).

Operative definitions:

1. Chest compression depth: defined as the maximum posterior deflection of the sternum prior to chest recoil. In order to be accurate a non-compressible surface must be beneath the patient. It is considered shallow is it is less than 50 mm and deep is greater than 60mm. Adequate chest compression depth is defined as being between 50-60 mm.
2. Chest compression rate: defined as the frequency of chest compressions per minute. It is considered slow if less than 100 chest compressions are performed per minute, and too fast if greater than 120 compressions are performed per minute. This rate will be calculated during 60 seconds intervals while chest compressions are provided. Adequate chest compression rate is defined as being between 100 and 120 compressions per minute.
3. Incomplete release of compressions/Recoil: defined as "leaning" phenomenon in which force is not completely removed during compressions. This is best reported by a simple binary measure: complete or incomplete (>2500g residual leaning force). Adequate recoil will be complete chest wall recoil.

Primary Outcome Measures: Proportion of healthcare providers who are accurate in their visual assessment of CPR quality.

Secondary Outcome Measures:

1. Proportion of healthcare practitioners who accurately report CPR quality from position in relation to the patient (head, side and foot of bed).
2. Proportion of healthcare practitioners accurately identifying CPR errors (rate, depth, recoil).

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric acute care healthcare providers: such as nurses, nurse practitioners, respiratory therapists, physicians, residents, fellows
2. Those who work in ER or ICU setting regularly or rotate through this setting
3. Basic Life Support (BLS), Pediatric Advanced Life Support (PALS) or Advanced Cardiac Life Support (ACLS) certification within the past two years

Exclusion Criteria:

1. Anyone who has participated previously in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Proportion of healthcare providers who are accurate in their visual assessment of CPR quality. | Data is anticipated to be presented 4 months after it is collected.

SECONDARY OUTCOMES:
Proportion of healthcare practitioners who accurately report CPR quality from position in relation to the patient (head, side and foot of bed). | Data is anticipated to be presented 4 months after data is collected.
Proportion of healthcare practitioners accurately identifying CPR errors (rate, depth, recoil). | Data is anticipated to be presented about 4 months after it is collected.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cheng, MD, FRCPC, Principal Investigator — University of Calgary
Locations (1):
- KidSim-Aspire Simulation Research Lab, Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Background] Sutton R, Niles D, Nysaether J et al. Quantitative Analysis of CPR quality during in-hospital resuscitation of older children and adolescents. Pediatrics. 2009; 124 : 1930-8. Sutton R, Maltese M, Niles D et al. Quantitative analysis of chest compression interruption during in-hospital resuscitation of older children and adolescents. Resuscitation 2009; 80:1259-1263. Atkins DL et al. Epidemiology and Outcomes From Out-of-Hospital Cardiac Arrest in Children: The Resuscitation Outcomes Consortium Epistry-Cardiac Arrest. Circulation. 2009;119:1484-91. Atkins DL, Everson-Stewart S, Sears GK, Daya M, Osmond MH, Warden CR, Berg RA. Epidemiology and outcomes from out-of-hospital cardiac arrest in children: the Resuscitation Outcomes Consortium Epistry-Cardiac Arrest. Circulation. 2009;119:1484-1491.
- [Derived] Jones A, Lin Y, Nettel-Aguirre A, Gilfoyle E, Cheng A. Visual assessment of CPR quality during pediatric cardiac arrest: does point of view matter? Resuscitation. 2015 May;90:50-5. doi: 10.1016/j.resuscitation.2015.01.036. Epub 2015 Feb 26. PMID 25727057